CLINICAL TRIAL: NCT06694987
Title: SCORE! Non-Physician Health Worker (NPHW) Implementation Protocol (SIP).
Acronym: SIP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sonia Anand (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor-Investigator, Sonia Anand, Associate Vice-President, Global Health Department, Professor of Epidemiology, Vascular Medicine Specialist, Principal Investigator, McMaster University
Organization: McMaster University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SCORE! - SIP
Record Dates: First submitted 2024-10-11; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Hypertension; Diabetes Mellitus; Dyslipidemia; Metabolic Syndrome
Keywords: Cardiovascular; Healthy active living; Newcomer; Non-Physician Health Worker
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Dyslipidemias; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental, one group, pre-post design study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Implementation group. (Experimental): The study is based on the HOPE-4 protocol, where trained individuals will support participants in adhering to healthy lifestyle recommendations and support their access to a family physician to follow up on care recommendations.
  The NPHWs will be allied health professionals (e.g., pharmacists, internationally trained physicians, physiotherapists, nurses). The team will train them on study goals, responsibilities, data management, and follow-up, based on the HOPE-4 training manual. Training will be given once at the beginning of their role and then once annually.
  The NPHW will support the participant, if needed, in contacting the family doctor and assisting to arrange a follow-up study. If required, the family doctor can contact the NPHW. If further discussion is required or there are questions regarding the study that require further discussion, the NPHW will contact the study physician to address these issues.
  Interventions: Other: Non-Physician Health Worker

INTERVENTIONS:
Other: Non-Physician Health Worker — NPHW will aid participants in accessing a family doctor if required. The family doctor will receive a letter from the study, with suggested medication, based on the HOPE-4 algorithm. The family doctor may decide not to prescribe the recommended treatment or give another treatment (medication). In such case, the participant will still be part of the study and family physician's decision and reason why will be recorded. Follow-up will occur as per the visit schedule. All participants will attend a 20-minute follow-up visits in person at 0, 6 and 12 months, and via telephone at 3 and 9 months.
  Participants will be assessed to determine if: i. the patient was assessed by their family physician, ii. the family doctor initiated recommended medication treatment(s), iii. they are adhering to the medications as prescribed, iv. they implemented what the NPHW has recommended about dietary and lifestyle changes, using the specific, measurable, achivable, relevant, time-bound (SMART) for goals.

SUMMARY:
This study is a substudy of the Strenghtening Community Roots (SCORE!) Cohort study. The investigators will look for people, enrolled in the SCORE! Cohort study, with abnormal results related to blood sugar and fat, as well as high blood pressure and heart disease risks. The investigaors will try to help the community improve sugar, fat and blood pressure through trained people who are not necessarily a medical doctor but have health-sciences-training backgrounds. These people are called Non-Physician Health Workers (NPHW), and they will be under the direction of a medical doctor and will be also in close communication with the participants and the medical doctor to improve their health. This will happen through a total of 12 months, having online and on-site visits, for follow-up.

DETAILED DESCRIPTION:
Rationale: The study has been created to help SCORE! Cohort participants with cardiovascular (CV) risk to receive medical guidance and adopt healthy lifestyle recommendations through NPHW under the direction of family physicians.

Objectives: To improve/maintain CV health (measured by blood pressure, glucose levels, lipids) through implementation of simplified treatment algorithm, connection to a NPWH and referrals to primary care physicians for pharmacological management, over 12 months.

Study Design: Implementation Study.

Population: All adults 18 years or older enrolled in the SCORE! Cohort who have the following uncontrolled CV risk factors: hypertension, elevated non-High density lipoprotein (HDL) cholesterol as per the Heart Outcomes Prevention Evaluation - 4 (HOPE-4) trial criteria, and/or elevated glucose as indicated by the random glucose level or the hemoglobin A1c (HbA1C) ≥ 6.5%.

Study procedures: Participants will be identified from the SCORE! Cohort study. If the participant has CV risk factors, they will be invited to the study. After the consent procedure, the NPHW will follow an algorithm validated in the HOPE-4 trial. There will be five follow-ups over 12 months.

Primary/Secondary outcomes: A change in Framingham Risk Score (FRS) after 12 months / A change in lipid panel, blood pressure, and glucose/HbA1c, medication adherence, smoking/tobacco cessation.

Data analysis: Descriptive and multivariate analysis will be conducted on the individual level. The overall participant population will be assessed for the proportion of participants with established cardiovascular disease (CVD), and in those without CVD, the proportion of individuals with CV risk factors and the percentage of people in low, moderate, and high FRS categories.

ELIGIBILITY:
Participants will be identified from the SCORE! Cohort study who have previously received a letter indicating their cardiovascular risk score.

They are eligible if:

Uncontrolled CV risk factors will be defined as follows:

* Blood pressure measurements: systolic ≥ 140 or diastolic BP ≥ 90 mm Hg;
* Non-HDL cholesterol > 2.66 mmol/L;
* Random plasma glucose of ≥ 11.1 mmol/L or HbA1c% ≥ 6.5%

Exclusion criteria include:

* Involvement in another study or program that would interfere with the study protocol,
* Known history of coronary artery disease or stroke;
* Severe co-morbid conditions with life expectancy < 1 year,
* Pregnancy or plans to become pregnant within 12 months;
* Other serious conditions or logistic factors likely to interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Framinghman risk score (FRS) | 12 months
  A change in Framingham Risk Score from baseline to 12 months. Values are estimated as risk percentages (the likelihood) to have a major adverse cardiovascular events (MACE) within the next 10 years.
  < 10 % = Low risk 10-20 % = Intermediate risk > 20 % = High risk

SECONDARY OUTCOMES:
HbA1c | 12 months
  Change in HbA1c for diabetic individuals.
HbA1c | 12 months
  Proportion of patients with an HbA1c less than 7.0 percent.
Blood pressure | 12 months
  Change in blood pressure (BP) in mm/Hg.
Blood pressure | 12 months
  Change in BP as:
  Proportion of participants with well-controlled BP from baseline to 12 defined as Systolic Blood Pressure (SBP) lower than 140 mmHg in non-diabetic individuals, and SBP lower than 130 mmHg in diabetic individuals.
Lipid panel | 12 months
  Change in low density lipoproteins (LDL) (mmol/L).
Lipid Panel | 12 months
  Change in HDL (mmol/L)
Lipid panel | 12 months.
  Change in total cholesterol (mmol/L).
Lipid panel | 12 months
  Change in triglycerides (mmol/L).
Lipid Panel | 12 months
  Proportion of participants with LDL in target from baseline at 12 months: defined as less than 2.0 mmol/L for individuals with diabetes or who are hypertensive and over the age of 60 or individuals with moderate to high FRS. For those with LDL lower than 5.0 mmol/L - reduction of 50 percent or less than 2.50 mmol/L as per CCS guidelines.
InterHEART Risk Score (IHRS) | 12 months
  Change in Interheart risk score (IHRS).
  Low risk (< or equal to 9) for adverse cardiac event Intermediate risk (10 to 15) for adverse cardiac event High risk (16 or higher) for adverse cardiac event
Tobacco | 12 months
  Proportion of individuals who reduced smoking.
Tabocco | 12 months
  Proportion of participants who quit smoking.
Implementation of the recommended tratment. | 12 months
  Proportion of physicians who implemented the recommended medical therapy, by the study.
Adherence to the NPHW's recommendations | 12 months
  Proportion of participants who implemented changes to healthy active living (HAL), recommended by the NPHW.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Anand, MD, PhD, Principal Investigator — McMaster University; Lita Cameron, MD, MSc, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
We currently dont have plans for sharing IPD. If this changes in the future, the consent form explains as follow:
  The participant's personal, identifiable data will not be shared with anyone except with the participant's consent or as required by the laws of the province of Ontario. All information that could identify the participant, such as name and phone number, will only be accessible to the study members who need this information to contact the participant for study purposes (e.g., invite the participant to activities). Before the investigators analyze the data collected, all identifying information will be removed. The de-identified data will be retained until it no longer hold scientific value. If the participant previously consented to sharing of data with other researchers or to data repositories in the main cohort study, data from this study will also be shared. If the participant no longer wish for this to occur the investigators will be notified.
  HiREB # 17633

REFERENCES:
- [Background] Schwalm JD, McCready T, Lopez-Jaramillo P, Yusoff K, Attaran A, Lamelas P, Camacho PA, Majid F, Bangdiwala SI, Thabane L, Islam S, McKee M, Yusuf S. A community-based comprehensive intervention to reduce cardiovascular risk in hypertension (HOPE 4): a cluster-randomised controlled trial. Lancet. 2019 Oct 5;394(10205):1231-1242. doi: 10.1016/S0140-6736(19)31949-X. Epub 2019 Sep 2. PMID 31488369